CLINICAL TRIAL: NCT02145091
Title: Effects of Psilocybin on Behavior, Psychology and Brain Function in Long-term Meditators
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NA_00047665-2
Record Dates: First submitted 2014-05-20; First posted 2014-05-22 (Estimated); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Healthy
Keywords: Psilocybin; Hallucinogens; Pharmacologic Actions; Central Nervous System Agents; Therapeutic Uses; Psychotropic Drugs
MeSH Terms: interventions — Lactose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- One all-day session (Experimental): Participants will complete on all-day study session with a moderately-high dose of psilocybin.
  Preparation will include two days of screening, and an additional 8 hours of session preparation over at least 2 days. Follow-up will consist of an interview and MRI scan one day after the all-day session, a questionnaire follow-up 2 months after the all-day session, and a final follow-up 12-18 months after the all-day session.
  Interventions: Drug: Moderately-high dose of psilocybin; Drug: Placebo
- Two all-day sessions (Experimental): Participants will complete two all-day study sessions, the first with placebo and the second with a moderately-high dose of psilocybin.
  Preparation will include two days of screening and 8 hours of session preparation over at least 2 days, before the first all-day session. Follow-up will consist of an interview and MRI scan one day after each all-day session, a questionnaire follow-up 2 months after each all-day session, and a final follow-up 12-18 months after the second all-day session.
  Interventions: Drug: Moderately-high dose of psilocybin; Drug: Placebo
- Three all-day sessions (Experimental): Participants will complete three all-day study sessions, the first two with placebo and the third with a moderately-high dose of psilocybin. The majority of participants (over 90%) will be assigned to either one or two all-day sessions. A small minority of participants (less than 10%) will be assigned to three all-day sessions.
  Preparation will include two days of screening and 8 hours of session preparation over at least 2 days, before the first all-day session. Follow-up will consist of an interview and MRI scan one day after each all-day session, a questionnaire follow-up 2 months after each all-day session, and a final follow-up 12-18 months after the third all-day session.
  Interventions: Drug: Moderately-high dose of psilocybin; Drug: Placebo
- MRI of the acute effects of psilocybin (Experimental): This is an optional arm consisting of two sessions where either placebo, a very-low dose of psilocybin, or a moderately-low dose of psilocybin will be administered. During each session, participants will undergo MRI scanning shortly after the administration of each dose. Study sessions may occur over one or two days. Participants who have previously completed an all-day session with psilocybin in this study will be eligible to volunteer for this arm.
  Interventions: Drug: Moderately-low dose of psilocybin; Drug: Very-low dose of psilocybin; Drug: Placebo

INTERVENTIONS:
Drug: Moderately-high dose of psilocybin — Oral dose of a moderately-high dose of psilocybin.
  Other Names: O-phosphoryl-4-hydroxy-N,N-dimethyltryptamine
  Arms: One all-day session; Three all-day sessions; Two all-day sessions
Drug: Moderately-low dose of psilocybin — Oral dose of a moderately-low dose of psilocybin.
  Other Names: O-phosphoryl-4-hydroxy-N,N-dimethyltryptamine
  Arms: MRI of the acute effects of psilocybin
Drug: Very-low dose of psilocybin — Oral dose of a very-low dose of psilocybin.
  Other Names: O-phosphoryl-4-hydroxy-N,N-dimethyltryptamine
  Arms: MRI of the acute effects of psilocybin
Drug: Placebo — An oral placebo (lactose pill).
  Other Names: Lactose

SUMMARY:
This is a double-blind placebo-controlled study investigating the acute and persisting effects of psilocybin on meditation, spirituality, health, well-being, prosocial attitudes, and brain functioning.

DETAILED DESCRIPTION:
This study will use questionnaires and functional magnetic resonance imaging (fMRI) to examine the acute and persisting effects of psilocybin on brain function, meditation, spirituality, and psychology. The majority of the study procedures -- including screening, preparatory meetings, placebo and psilocybin sessions, and a large battery of behavioral and psychological measures -- will be conducted at the investigator's laboratory at the Behavioral Pharmacology Research Unit (BPRU) on the Johns Hopkins Bayview campus. The brain imaging procedures will be conducted at F.M. Kirby Research Center at the Kennedy Krieger Institute (KKI).

ELIGIBILITY:
Inclusion criteria:

* Have given written informed consent
* Some college-level education (college degree preferred)
* Be healthy and psychologically stable as determined by screening for medical and psychiatric problems via a personal interview, a medical questionnaire, a physical examination, an electrocardiogram (ECG), and routine medical blood and urinalysis laboratory tests
* Agree to consume approximately the same amount of caffeine-containing beverage (e.g., coffee, tea) that he/she consumes on a usual morning, before arriving at the research unit on the mornings of drug session days. If the participant does not routinely consume caffeinated beverages, he/she must agree not to do so on session days.
* Agree to refrain from using any psychoactive drugs, including alcoholic beverages and nicotine, within 24 hours of each drug administration. The exception is caffeine. Participants will be required to be non-smokers.
* Agree not to take any Pro re-nata (PRN) medications on the mornings of drug sessions
* Agree not to take sildenafil (Viagra®), tadalafil, or similar medications within 72 hours of each drug administration.
* Agree that for one week before each drug session, he/she will refrain from taking any nonprescription medication, nutritional supplement, or herbal supplement except when approved by the study investigators. Exceptions will be evaluated by the study investigators and will include acetaminophen, non-steroidal anti-inflammatory drugs, and common doses of vitamins and minerals.
* Live within driving distance of Baltimore - out-of-State residents may be eligible if they can provide their own transportation and lodging.
* Have a long-term meditation practice, ideally in a Buddhist tradition, with good familiarity with breath meditation and loving kindness meditation; preference given to those with very long-term practices

Exclusion criteria:

* Women who are pregnant (as indicated by a positive urine pregnancy test assessed at intake and before each drug session) or nursing; women who are of child-bearing potential and sexually active who are not practicing an effective means of birth control.
* Cardiovascular conditions: coronary artery disease, stroke, angina, uncontrolled hypertension, a clinically significant ECG abnormality (e.g., atrial fibrilation), or Transient Ischemic Attack (TIA) in the past year
* Epilepsy with history of seizures
* Insulin-dependent diabetes; if taking oral hypoglycemic agent, then no history of hypoglycemia
* Currently taking psychoactive prescription medication on a regular (e.g., daily) basis
* Currently taking on a regular (e.g., daily) basis any medications having a primary centrally-acting pharmacological effect on serotonin neurons or medications that are Monoamine Oxidase (MAO) inhibitors. For individuals who have intermittent or PRN use of such medications, psilocybin sessions will not be conducted until at least 5 half-lives of the agent have elapsed after the last dose.
* More than 20% outside the upper or lower range of ideal body weight according to Metropolitan Life height and weight table
* Head trauma
* Claustrophobia
* Cardiac pacemaker
* Implanted cardiac defibrillator
* Aneurysm brain clip
* Inner ear implant
* Artificial heart valve (last 6 weeks)
* Prior history as a metal worker and/or certain metallic objects in the body

Psychiatric Exclusion Criteria:

* Current or past history of meeting Diagnostic and Statistical Manual (DSM)-IV criteria for Schizophrenia, Psychotic Disorder (unless substance-induced or due to a medical condition), or Bipolar I or II Disorder
* Current or past history within the last 5 years of meeting DSM-IV criteria for alcohol or drug dependence (excluding caffeine and nicotine) or severe major depression
* Have a first or second-degree relative with Schizophrenia, Psychotic Disorder (unless substance induced or due to a medical condition), or Bipolar I or II Disorder
* Has a psychiatric condition judged to be incompatible with establishment of rapport or safe exposure to psilocybin

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-05; Primary Completion 2019-12-26 (Actual); Study Completion 2019-12-26 (Actual)

PRIMARY OUTCOMES:
Persisting Effects Questionnaire | 2 months and 12-18 months post-session
  This is a measure of changes in spirituality, personal well-being, relationships, and emotions.
Hood Mysticism Scale | End of session day.
  This measures subjective experiences associated with classical mystical experiences.
States of Consciousness Questionnaire | End of session day
  Measures subjective experience associated with classical mystical experiences.
fMRI Resting State Functional Connectivity | 2 months pre and 1 day post session
  Measures change in activity in brain regions that have been previously shown to be modulated by either psilocybin or meditation.

CONTACTS AND LOCATIONS:
Locations (1):
- Behavioral Pharmacology Research Unit, Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States